CLINICAL TRIAL: NCT03514745
Title: Comparison of Lighted Stylet and GlideScope for Double-lumen Endobronchial Intubation in Patients With a Predicted Difficult Airway
Brief Title: Comparison of Lighted Stylet and GlideScope for Double-lumen Endobronchial Intubation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jin-Young Hwang, MD.PhD., SMG-SNU Boramae Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 20171227
Record Dates: First submitted 2018-04-20; First posted 2018-05-02 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Intubation;Difficult

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GlideScope group (Active Comparator): After the induction of anesthesia, endobronchial intubation is performed using the GlideScope.
  Interventions: Device: GlideScope
- Lighted stylet group (Experimental): After the induction of anesthesia, endobronchial intubation is performed using a lighted stylet.
  Interventions: Device: Lighted stylet

INTERVENTIONS:
Device: GlideScope — Endobronchial intubation is performed using the GlideScope.
  Arms: GlideScope group
Device: Lighted stylet — Endobronchial intubation is performed using a lighted stylet.
  Arms: Lighted stylet group

SUMMARY:
We evaluate the GlideScope and lighted stylet for DLT intubation in terms of the intubation time, number of intubation attempts, difficulty in DLT advancement towards the glottis, postoperative sore throat and hoarseness, and hemodynamic responses during intubation in patients with predicted difficult airways.

ELIGIBILITY:
Inclusion Criteria:

* adult patients undergoing thoracic surgery requiring endobronchial intubation for one-lung ventilation

Exclusion Criteria:

* presence of sore throat and hoarseness
* requirements for postoperative mechanical ventilation
* at risk of aspiration.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-05-06 (Actual); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Intubation time taken for endobronchial intubation | During endobronchial intubation
  Intubation time is defined as the time elapsed from picking up GlideScope or lighted stylet to confirmation of successful intubation by capnometry.

SECONDARY OUTCOMES:
Number of intubation attempts | During endobronchial intubation
  Total intubation attempts are counted.
Difficulty of DLT advancement towards the glottis | During endobronchial intubation
  It is categorised as very easy, easy, difficult, and very difficult
Resistance to DLT insertion through the glottis | During endobronchial intubation
  It is categorized as none, mild, and moderate
The incidence and severity of postoperative sore throat | At 1 and 24 hours after surgery
  It is quantified by using a 100-point numerical rating scale (NRS, 0 [no pain], 100 [worst pain imaginable]).
The incidence and severity of postoperative hoarseness | At 1 and 24 hours after surgery
  Hoarseness is defined as a voice quality different from the preoperative voice and graded as follows: none (no hoarseness), mild (recognized by the patient), moderate (obvious to the investigator), and severe (aphonia).

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Young Hwang, M.D., Ph.D., Study Director — Seoul Metropolitan Government Seoup National University Boramae Medical Center
Locations (1):
- Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul, South Korea